CLINICAL TRIAL: NCT06604559
Title: The Effect of Patient Discharge From the Maternal and Fetal Medicine Unit With Receiving a Discharge Letter Later Using the Apollo App on Discharge Data, Safety and Patient Satisfaction - a Prospective Randomized Controlled Trial
Brief Title: The Effect of Patient Discharge From the Maternal and Fetal Medicine Unit With Receiving a Discharge Letter Later Using the Apollo App on Discharge Data, Safety and Patient Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 55-24-POR
Record Dates: First submitted 2024-08-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Patient Satisfaction; Health Care Utilization
MeSH Terms: conditions — Patient Satisfaction; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application discharge (Experimental): The discharge is conditional on the approval of a senior physician or the attending physician in charge. The participant will sign on a "Form for discharge and consent to receive a discharge letter, using the "Apollo" application" in which the discharge process, recommendations and contact information of the department are described. Thereafter, the patient will be discharge home and the discharge letter will be available in the app once it is written. The participant is guided to contact the department, in case the discharge letter is not received in the application up to 24 hours after discharge.
  Interventions: Other: Discharge using Apollo application
- Regular discharge (Other): The discharge is conditional on the approval of a senior physician or the attending physician in charge. The patient will go home only after the discharge letter is written.
  Interventions: Other: Regular discharge

INTERVENTIONS:
Other: Discharge using Apollo application — Discharge using Apollo application
  Arms: Application discharge
Other: Regular discharge — Discharge with the regular process
  Arms: Regular discharge

SUMMARY:
Women admitted to the maternal and fetal medicine unit are often discharged after a short hospital stay. The routine work in the department is prioritized such that the discharge letter are written. In the last year the Apollo mobile application (app) was introduced. It contains general information on the medical center and the maternal and fetal unit department as well as the medical records, laboratory results and summary and discharge letters. The Apollo app is used in the maternal and fetal unit in the discharge process so the patient can receive the discharge letter in the app and does not need to wait until the discharge letter is written.

It is not known whether this process is more effective than the regular discharge process and patients' satisfaction was not assessed previously.

In the present study we will compare discharge data, satisfaction and safety of discharging using the Apollo app versus the routine process.

ELIGIBILITY:
Inclusion Criteria:

* Women who are admitted to the maternal and fetal medicine unit with the intention to be discharged before delivery
* 18 years old and older
* Consent to participate
* Owner of a smart phone
* Consent to download the Apollo app

Exclusion Criteria:

* Delivery during her admission
* Doesn't own a smart phone
* Refusal to download to Apollo app
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
The mean time needed from discharge decision until the actual discharge | up to 24 hours from discharge decision

SECONDARY OUTCOMES:
Satisfaction rate from the discharge method | Within a week following discharge from the department
  Satisfaction rate from the discharge method assessment using a questionnaire
The rate of participants with any technical difficulties to receive the discharge letter and reasons | Within a week following discharge from the department using a questionnaire
  The rate of participants with any technical difficulties to receive the discharge letter and reasons using a questionnaire
The rate of participants with missed information that required the patient to seek medical help | Within a week following discharge from the department using a questionnaire
  The rate of participants with missed information that required the patient to seek medical help using a questionnaire
The rate of participants with discrepancies between the discharge recommendations written in the final discharge letter and the "Form for discharge and consent to receive a discharge letter, using application" and details regarding the discripancies | Within a week following discharge from the department

CONTACTS AND LOCATIONS:
Locations (1):
- Tzafon Medical center, Poriya, Tiberias, North, Israel

IPD SHARING:
Plan to Share IPD: No